CLINICAL TRIAL: NCT01201291
Title: Impact of Inspired Oxygen Fraction on Outcome in Patients With Traumatic Brain Injury
Acronym: BRAINOXY
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to slow recruitment the study was terminated
Sponsor: Kuopio University Hospital (Other)
Collaborators: Tampere University Hospital (Other); Turku University Hospital (Other Government); Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Stepani Bendel, MD, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KUH5070218
Record Dates: First submitted 2010-09-13; First posted 2010-09-14 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Traumatic Brain Injury | Patient
Keywords: TBI; Normobaric hyperoxia; Outcome; GOS; GOSE

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fraction of inspired oxygen of 0.4 (Active Comparator): Fraction of inspired normobaric oxygen of 0.4 (low oxygen group)
  Interventions: Other: Normobaric oxygen
- Fraction of inspired oxygen of 0.7 (Active Comparator): Fraction of inspired normobaric oxygen of 0.7 (high oxygen group)
  Interventions: Other: Normobaric oxygen

INTERVENTIONS:
Other: Normobaric oxygen — Fraction of inspired oxygen

SUMMARY:
Aim of the study is to investigate the impact of two different fractions of inspired oxygen (FiO2) on outcome in patients with severe traumatic brain injury (TBI).

DETAILED DESCRIPTION:
The high oxygen group is treated during mechanical ventilation with either a fraction of inspired oxygen of 0.7 (high oxygen group) or a fraction of inspired oxygen 0.4 (control group). The intervention continues until withdrawal of mechanical ventilation, ICU discharge or until 14 days from ICU randomisation.

Primary outcome is worse than expected outcome in the corresponding treatment arms based on outcome meas-ured by the probability of bad outcome using the CRASH® risk calculator (prognostic model for predicting outcome after traumatic brain injury).

Secondary outcome is occurence of lung injury during mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with isolated non-penetrating traumatic brain injury
* Multiple trauma patient with brain injury and traumas outside abdomen, thorax or pelvis not affecting oxygenation
* Glasgow coma scale eight or less (inclusive)
* Expected need for intubation and for mechanical ventilation more than 24 hours.
* Are recruited <18 hours after admittance to ICU and
* Time from TBI is less than 36 hours
* Informed consent from patients representative

Exclusion Criteria:

* Age <18 or >65 years,
* Anticipated brain death in 12 hours (donor treatment) or otherwise moribund patient expected to die in 24 hours
* Expected need for mechanical ventilation less than 24 hours
* Insufficient oxygenation assessed by a clinician or multiple trauma patients with brain injury and severe abdominal, thoracic or pelvic injury possibly affecting oxygenation.
* No consent
* Insufficient oxygenation with the treatment modality of the lower oxygenation group (Pa02 less than 13 kPa or SpO2 95% with Fi02 40%, PEEP 10 or less) or oxygenation failure probable during ICU care (severe aspiration, multiple trauma patients with brain injury and severe abdominal, thoracic or pelvic injury possibly affecting oxygenation)
* Penetrating TBI
* No consent
* Suspected pregnancy (perform urinary or serological pregnancy test if suspected)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2010-11; Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Glasgow outcome scale(GOS) and/or Extended glasgow outcome scale (GOSE) | 6 months
  The study is powered to have 80% power at 5% significance level to detect a treatment effect that decreases the proportion of poor outcome from 55% to 45%.
  Each patient is given an individualized tailored prognosis based on patient's baseline prognosis in a large reference population. Outcome is measured by using functional outcome score, Glasgow outcome score (GOS) and/or GOS extended (GOSE).

SECONDARY OUTCOMES:
6 month outcome | 6 months
  Combined proportion of unfavourable neurological outcomes at 6 months:
  severe disability (GOSE 2-4) or death (GOSE 1):
  Occurence of lung injury during mechanical ventilation: ALI-criteria or ARDS criteria used (paO2/FiO2 ratio less than 300 or 200 respectively):
  Mortality at 6 months:
  Proportion of surviving patients with unfavourable neurological outcome at 6 months (GOSE 2-4).
  Quality of life assessment (EQ-5D) at 6 months:
  Prolonged mechanical ventilation Re-intubation rates

CONTACTS AND LOCATIONS:
Overall Officials: Esko Ruokonen, Professor, Principal Investigator — Kuopio University Hospital; Stepani J Bendel, MD,PhD, Study Director — Kuopio University Hospital; Maarit Lång, MD, Principal Investigator — Kuopio University Hospital
Locations (4):
- Finland (4):
  - Helsinki University Central Hospital, Töölö Hospital, Helsinki, Töölö
  - Kuopio University Hospital, Kuopio
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku

IPD SHARING:
Plan to Share IPD: Undecided